CLINICAL TRIAL: NCT03051698
Title: Effect of Intravenous Administration of C1-inhibitor on Inflammation and Coagulation After Bronchial Instillation of House Dust Mite Allergen and Lipopolysaccharide in Allergic Asthma Patients
Brief Title: C1-inhibitor in Allergic ASThma Patients
Acronym: CAST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed no differences between groups
Sponsor: T. van der Poll (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Prothya Biosolutions (Industry)
Responsible Party: Sponsor-Investigator, T. van der Poll, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015_024
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Asthma
Keywords: C1-inhibitor; house dust mite; complement system
MeSH Terms: conditions — Asthma; Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein; SERPING1 protein, human; Sodium Chloride; Anti-Bacterial Agents; Vancomycin; Ciprofloxacin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- C1-inhibitor (Experimental): One gift of intravenous administration of C1-inhibitor (Cinryze, 100U/kg) during one hour
  Interventions: Drug: C1-inhibitor
- Saline (Placebo Comparator): One gift of intravenous administration of 0.9% NaCl during one hour.
  Interventions: Other: Saline
- Antibiotics (Experimental): broad spectrum antibiotics (vancomycin, ciprofloxacin, metronidazole) for 7 days (washout 36 hours before study day).
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: C1-inhibitor — 100 Unit/kg IV, one gift prior to broncho provocation.
  Other Names: Cinryze
  Arms: C1-inhibitor
Other: Saline — 0.9% NaCl
  Arms: Saline
Drug: Antibiotics — vancomycin, ciprofloxacin, metronidazole
  Other Names: vancomycin, ciprofloxacin, metronidazole
  Arms: Antibiotics

SUMMARY:
The purpose of this proof-of-concept study is to determine the effect of Intestinal Microbiota Depletion or Intravenous Administration of C1-inhibitor on Inflammation and Coagulation after Bronchial Instillation of House Dust Mite Allergen and Lipopolysaccharide in Allergic Asthma Patients

DETAILED DESCRIPTION:
Intravenous administration of C1-inhibitor (n=20) or vehicle (n=20). One group of patients (n=20) will receive broad spectrum antibiotics (vancomycin, ciprofloxacin, metronidazole) for 7 days (washout 36 hours before study day). This group will receive the same vehicle as the control group 2 hours prior to challenge. HDM will be administered together with the environmental pollutant LPS in a lung subsegment via a bronchoscope (mimicking environmental exposure to HDM); a contralateral lung subsegment will be administered with saline (control side). After 7 hours, bronchoalveolar lavage (BAL) fluid will be harvested by a second bronchoscopy. Blood samples will be collected before administration of C1-inhibitor or vehicle, and before both bronchoscopies. Faeces will be collected prior to antibiotic administration as well as prior to HDM+LPS challenge.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent to mild asthma according to the Global Initiative for Asthma (GINA) criteria
* Allergy for HDM documented by a positive RAST and a positive skin prick test.
* No clinically significant findings during physical examination and hematological and biochemical screening
* At spirometry FEV1 more than 70% of predicted value
* A PC20 between 0.3 - 9.6 mg/ml (corresponding with increased airway hyperreactivity)
* Able to communicate well with the investigator and to comply with the requirements of the study
* Stable asthma without the use of asthma medication 2 weeks prior to the study day. As documented by the Juniper's Asthma control questionnaire (ACQ) score < 1,2.
* Written informed consent
* No current smoking for at least 1 year and less than 10 pack years of smoking history

Exclusion Criteria:

* Relevant comorbidity, pregnancy and/or recent surgical procedures.
* A history of smoking within the last 12 months, or regular consumption of greater than three units of alcohol per day
* Exacerbation and/ or the use of asthma medication within 2 weeks before start
* Administration of any investigational drug within 30 days of study initiation
* Donation of blood within 60 days, or loss of greater than 400 ml of blood within 12 weeks of study initiation]
* History of venous or arterial thromboembolic disease
* History of enhanced bleeding tendency or abnormal clotting test results.
* History of serious drug-related reactions, including hypersensitivity
* Inability to maintain stable without the use of asthma medication 2 weeks before start of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Influx of inflammatory cells in the lung | 7 hours after bronchial instillation of house dust mite (HDM) and lipopolyssacharide(LPS)
  Most important cell types are the eosinophils and neutrophils in bronchoaveolar fluid

SECONDARY OUTCOMES:
Interleukin-4 in pg/ml. | 7 hours after bronchial instillation of HDM and LPS
Interleukin-5 in pg/ml. | 7 hours after bronchial instillation of HDM and LPS
IL-13 in pg/ml. | 7 hours after bronchial instillation of HDM and LPS
IL-10 in pg/ml. | 7 hours after bronchial instillation of HDM and LPS
IFN-Y in pg/ml. | 7 hours after bronchial instillation of HDM and LPS
TNF-α in pg/ml. | 7 hours after bronchial instillation of HDM and LPS
CCL11 in pg/ml. | 7 hours after bronchial instillation of HDM and LPS
Interleukin-6 in pg/ml. | 7 hours after bronchial instillation of HDM and LPS
C4bc u/ml | 7 hours after bronchial instillation of HDM and LPS
C3bc u/ml | 7 hours after bronchial instillation of HDM and LPS
iC3b u/ml | 7 hours after bronchial instillation of HDM and LPS
C5a ng/ml | 7 hours after bronchial instillation of HDM and LPS
C5b-9 u/ml. | 7 hours after bronchial instillation of HDM and LPS
C3a in ng/ml | 7 hours after bronchial instillation of HDM and LPS
FXIIa activity in OD | 7 hours after bronchial instillation of HDM and LPS
FXIa in OD | 7 hours after bronchial instillation of HDM and LPS
FXIIa- C1-inhibitor complexes u/ml | 7 hours after bronchial instillation of HDM and LPS
kallikrein-C1-inhibitor complexes u/ml | 7 hours after bronchial instillation of HDM and LPS
high-molecular weight kininogen in AU | 7 hours after bronchial instillation of HDM and LPS
thrombin-antithrombin complexes in ng/ml. | 7 hours after bronchial instillation of HDM and LPS

OTHER OUTCOMES:
C1-inhibitor activity in bronchoalveolar lavage | 7 hours after bronchial instillation of HDM and LPS

CONTACTS AND LOCATIONS:
Overall Officials: Tom vd Poll, Prof, dr, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeerleder S. C1-inhibitor: more than a serine protease inhibitor. Semin Thromb Hemost. 2011 Jun;37(4):362-74. doi: 10.1055/s-0031-1276585. Epub 2011 Jul 30. PMID 21805442
- [Background] Zhang X, Kohl J. A complex role for complement in allergic asthma. Expert Rev Clin Immunol. 2010 Mar;6(2):269-77. doi: 10.1586/eci.09.84. PMID 20402389
- [Background] Schmudde I, Laumonnier Y, Kohl J. Anaphylatoxins coordinate innate and adaptive immune responses in allergic asthma. Semin Immunol. 2013 Feb;25(1):2-11. doi: 10.1016/j.smim.2013.04.009. Epub 2013 May 19. PMID 23694705
- [Background] de Boer JD, Berger M, Majoor CJ, Kager LM, Meijers JC, Terpstra S, Nieuwland R, Boing AN, Lutter R, Wouters D, van Mierlo GJ, Zeerleder SS, Bel EH, van't Veer C, de Vos AF, van der Zee JS, van der Poll T. Activated protein C inhibits neutrophil migration in allergic asthma: a randomised trial. Eur Respir J. 2015 Dec;46(6):1636-44. doi: 10.1183/13993003.00459-2015. Epub 2015 Sep 17. PMID 26381519
- [Background] Bel EH. Mild asthma. N Engl J Med. 2013 Dec 12;369(24):2362. doi: 10.1056/NEJMc1313111. No abstract available. PMID 24328483
- [Background] Krug N, Tschernig T, Erpenbeck VJ, Hohlfeld JM, Kohl J. Complement factors C3a and C5a are increased in bronchoalveolar lavage fluid after segmental allergen provocation in subjects with asthma. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1841-3. doi: 10.1164/ajrccm.164.10.2010096. PMID 11734433
- [Derived] Van Engelen TSR, Yang J, Haak BW, Bonta PI, Van Der Poll T, Wiersinga WJ; CAST study group. Gut Microbiome Modulation by Antibiotics in Adult Asthma: A Human Proof-of-Concept Intervention Trial. Clin Gastroenterol Hepatol. 2022 Jun;20(6):1404-1407.e4. doi: 10.1016/j.cgh.2021.07.030. Epub 2021 Jul 22. PMID 34303860